CLINICAL TRIAL: NCT04864808
Title: Treating ADHD Parents and Their Infants Via Telehealth: Developing an Early Parenting Intervention Using a Deployment-focused Intervention Design
Brief Title: Helping Toddlers and Parents Together
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Qualitative interviews were conducted with stakeholders and informed the intervention development. However, due to professional and personal medical reasons, the PI was given permission by NIH to discontinue the case series.
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Andrea Chronis-Tuscano, Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH118320-02S1 (NIH); R01MH118320-02S1 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-04-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: ADHD; Parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Parenting Training (Experimental)
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Parents will receive sessions of behavioral parent training with components specifically targeted toward parents with ADHD. The number of sessions will be informed based on stakeholder feedback. Treatment will be delivered via telehealth.

SUMMARY:
Using stakeholder feedback (i.e., behavioral health providers & caregivers), the goal of this study is to develop a behavioral parenting program that focuses on both parent mental health and parenting for parents of toddlers (12-35 months old). Using a deployment focused intervention model, this study will : (1) develop an early parenting intervention for parents of at-risk toddlers which integrates a focus on parent mental health with evidence-based behavioral parenting strategies, and (2) examine context-specific factors related to the intervention, including feasibility and acceptability to design a more practice-ready intervention.

DETAILED DESCRIPTION:
Very early identification of children and families at risk of developing psychopathology can lead to early prevention/intervention to address challenging behaviors before they become more severe, likely reducing the length and cost of interventions. Using the information provided by the stakeholder group, the current study will implement in an open trial the early parenting intervention for ADHD parents of at-risk toddlers (n = 10 families) via telehealth by primary care co-located psychologists. Investigators will examine implementation factors including fidelity, feasibility (utility, adherence) and acceptability (facilitators, barriers) of the early parenting intervention. Quantitative data (adherence checklists, symptom measures, observational parenting measures) will be used to assess the extent to which primary care providers and office staff adhere to the intervention manual, as well as changes in toddler and parent behavior resulting from the intervention. Qualitative data (interviews/ focus groups) with stakeholders (behavioral health providers and caregivers of toddlers) will inform a refined intervention model and assess perceptions of utility, fit, and satisfaction of the intervention components. This mixed-methods approach will offer the most comprehensive examination of an early parenting intervention model for parents of at-risk toddlers in a pediatric primary care setting.

ELIGIBILITY:
Inclusion Criteria:

- To be included in the stakeholder group, participants must work at a CNMC primary center or must be a parent with a toddler.

For inclusion to participate in the pilot intervention, a full-time guardian must, at the time of screening:

1. Sign informed consent online
2. Be between 21-55 years old (inclusive) and be English or Spanish-speaking
3. Meet full DSM-5 criteria for ADHD, any subtype as determined by the SCID-5
4. Have current CGI-S-ADHD rating ≥ 4 and < 7
5. Commit to the entire study
6. Be able to complete all study assessments virtually (i.e., they must have a device that connects to the internet with a camera)

Parents with common comorbid conditions will be included provided that: (a) they do not report active suicidal ideation with intent; and (b) if receiving an antidepressant medication, their medication is well-tolerated and has not changed within 30 days.

For inclusion to participate in the pilot intervention, toddlers must:

1. be between ages of 12 - 35 months at time of consent
2. score above the 75th percentile on the BITSEA problem scale

Exclusion Criteria:

* Parents will be excluded on the basis of current bipolar disorder, schizophrenia, psychoses, or other primary psychiatric disorder requiring other immediate treatment.

Ages: 12 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Acceptability | up to 12 weeks
  Client Satisfaction Questionnaire (CSQ-8)- higher scores indicate more satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Chronis-Tuscano, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chronis-Tuscano A, O'Brien KA, Johnston C, Jones HA, Clarke TL, Raggi VL, Rooney ME, Diaz Y, Pian J, Seymour KE. The relation between maternal ADHD symptoms & improvement in child behavior following brief behavioral parent training is mediated by change in negative parenting. J Abnorm Child Psychol. 2011 Oct;39(7):1047-57. doi: 10.1007/s10802-011-9518-2. PMID 21537894
- [Background] Bagner DM, Coxe S, Hungerford GM, Garcia D, Barroso NE, Hernandez J, Rosa-Olivares J. Behavioral Parent Training in Infancy: A Window of Opportunity for High-Risk Families. J Abnorm Child Psychol. 2016 Jul;44(5):901-12. doi: 10.1007/s10802-015-0089-5. PMID 26446726